CLINICAL TRIAL: NCT06906419
Title: Evaluering av Kliniske Resultater Hos Pasienter Operert for Kronisk Residiverende Patellaluksasjoner Ved Hjelp av Artroskopisk Stabilisering Med Trokleaplastikk. En Kvalitetskontroll-studie
Brief Title: Arthroscopic Trochleaplasty in Chronic Relapsing Patellar Dislocations: A Follow-up Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1000324
Record Dates: First submitted 2025-03-07; First posted 2025-04-02 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Patellar Dislocation
Keywords: patellar dislocation; arthroscopic; trochleaplasty
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the long-term clinical outcomes of arthroscopic trochleoplasty in patients treated for chronic recurrent patellar dislocations. The primary objective is to assess the effectiveness of the procedure in reducing the need for re-operations and preventing recurrent instability. Secondary objectives include evaluating postoperative complications, patellofemoral pain, functional outcomes using the Kujala Anterior Knee Pain Scale (AKPS), and quality of life measured by EQ-5D-5L. This retrospective cohort study will analyze data from patient records and structured telephone interviews conducted at least one year post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Underwent arthroscopic trochleoplasty for chronic recurrent patellar dislocations.
* Surgery performed between 2015 and 2023.
* Availability of follow-up data and consent for participation.

Exclusion Criteria:

* Concurrent knee surgeries unrelated to trochleoplasty.
* Previous surgeries on the same knee.
* Other significant orthopedic conditions affecting the knee.
* Lack of follow-up data or consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study evaluates the long-term outcomes of arthroscopic trochleoplasty performed to stabilize the patella in patients with chronic recurrent dislocations. The procedure involves deepening the trochlea femoris to enhance patellar tracking and prevent lateral dislocation. In some cases, medial patellofemoral ligament (MPFL) reconstruction was also performed. Data will be collected through patient medical records and structured telephone interviews, focusing on re-operation rates, postoperative complications, pain levels, functional outcomes, and quality of life. The study seeks to provide insights into the effectiveness and safety of this surgical technique, aiming to optimize treatment protocols for patellar instability.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Re-operation Rate | The investigators seek to register any re-operations from the time between the index surgery and the interview, ranging from 1 year up to 7 years postoperatively.
  Proportion of patients requiring additional surgical interventions after the index surgery at our institution.

SECONDARY OUTCOMES:
Recurrent Instability Rate | The investigators seek to register any incidences of recurrent instability from the time between the index surgery and the interview, ranging from 1 year up to 7 years postoperatively.
  Incidence of recurrent patellar dislocations post-surgery.
Postoperative Complications | The investigators seek to register any complications related to the index surgery from the time between the index surgery and the interview, ranging from 1 year up to 7 years postoperatively.
  Frequency and type of complications following trochleoplasty.
Functional Outcome | At the time of the interview, which will be performed from 1 year up to 7 years postoperatively.
  Kujala Anterior Knee Pain Scale (AKPS) scores assessing pain and knee function. The Kujala Score or Anterior Knee Pain Scale (AKPS) is a 13-item self-report questionnaire that assesses subjective reactions to particular activities and symptoms that are known to correlate with anterior knee pain syndrome. The AKPS is graded on a scale of 0 to 100, with 100 being the highest possible score. Lower scores reflect greater pain and disability.
EQ-5D-5L (HRQoL) scores | At the time of the follow-up interview, which will be performed from 1 year up to 7 years postoperatively.
  EQ-5D-5L (HRQoL) scores evaluating general health and well-being. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Pain Assessment | At the time of the follow-up interview, which will be performed from 1 year up to 7 years postoperatively.
  Numeric pain rating scale (NRS), ranging from the least pain, 0, to the worst pain imaginable, 10, during daily activities.
Patient Satisfaction | At the time of the follow-up interview, which will be performed from 1 year up to 7 years postoperatively.
  Satisfaction score on a scale, ranging from 1 (very dissatisfied) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Vestre Viken HF, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No